CLINICAL TRIAL: NCT05505669
Title: Circulating Biomarkers of Beta Cell Loss/Dysfunction in Diabetes
Brief Title: Circulating Biomarkers in the Development of Type 1 Diabetes
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20477; R01DK125856 (NIH)
Record Dates: First submitted 2022-07-31; First posted 2022-08-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urinary, saliva, plasma and serum samples are collected for future analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Adults with type 1 diabetes: Adults with type 1 diabetes
  Interventions: Other: One-time blood (up to 100 ml) will be drawn and the amount of blood drawn is based on weight. Saliva and urine will be collected during the blood draw visit.
- Adult healthy volunteers: Adult healthy volunteers
  Interventions: Other: One-time blood (up to 100 ml) will be drawn and the amount of blood drawn is based on weight. Saliva and urine will be collected during the blood draw visit.
- Children with type 1 diabetes: Children with type 1 diabetes
  Interventions: Other: One-time blood (up to 100 ml) will be drawn and the amount of blood drawn is based on weight. Saliva and urine will be collected during the blood draw visit.
- Adults with type 2 diabetes: Adults with type 2 diabetes
  Interventions: Other: One-time blood (up to 100 ml) will be drawn and the amount of blood drawn is based on weight. Saliva and urine will be collected during the blood draw visit.
- Adults with high blood sugar: Adults with high blood sugar
  Interventions: Other: One-time blood (up to 100 ml) will be drawn and the amount of blood drawn is based on weight. Saliva and urine will be collected during the blood draw visit.
- Those at risk of developing type 1 diabetes: Those at risk of developing type 1 diabetes
  Interventions: Other: One-time blood (up to 100 ml) will be drawn and the amount of blood drawn is based on weight. Saliva and urine will be collected during the blood draw visit.

INTERVENTIONS:
Other: One-time blood (up to 100 ml) will be drawn and the amount of blood drawn is based on weight. Saliva and urine will be collected during the blood draw visit. — One-time blood (up to 100 ml) will be drawn and the amount of blood drawn is based on weight. Saliva and urine will be collected during the blood draw visit.

SUMMARY:
More than 100 million U.S. adults are now living with diabetes or prediabetes. Investigators still do not fully understand how diabetes develops and how the disease worsens. Insulin is a hormone that helps the body use sugar as a fuel and control blood-sugar levels. People with diabetes have problems making insulin. This is because their insulin-producing beta cells -in the pancreas-are damaged or destroyed. A biomarker is a biological molecule (such as DNA, RNA (the genetic material of cells) or protein) that is a sign of a normal or abnormal process, or of a condition or disease. A biomarker can be measured and found in blood and/or other body fluids (such as saliva and urine). Understanding the biology of beta cells could help find diabetes-related biomarkers. The discoveries from this research could help with early diagnosis of diabetes and lead to the creation of therapies for treating diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent/ assent from the subject
* ONE of the following:

  * Type 1 diabetes patients (including pediatric patients) -OR-
  * Adult type 2 diabetes patients -OR-
  * Volunteers who are islet auto-antibody positive (i.e. insulin, GAA, IA-2, IAA and ZnT8 antibodies) with HbA1c ≤ 5.6% (including pediatric patients)-OR-
  * Adult participants with clinical diagnosis of high blood sugar (i.e. HbA1c of 5.7% to 6.4%)-OR-
  * Adult control subjects with HbA1cc ≤ 5.6%
* Weight ≥ 30 kg
* Willingness to: Provide blood sample(s) and if applicable: permit medical record/ clinical laboratory result review

Exclusion Criteria:

* Control subjects must not have any chronic conditions or have undergone cellular, tissue or organ transplant
* Sickle cell disease or anemia (exception: anemia that is corrected with treatment and source documents confirm corrected blood parameters current within 6 months of blood draw)
* Active infection
* Active malignancy (i.e., currently undergoing treatment)
* Immunomodulatory therapy within 1 year of planned blood draw (may include immune checkpoint inhibitors, thalidomide, lenalidomide, pomalidomide, imiquimod, Bacillus Calmette-Guérin, and cytokines/ growth factors (e.g. interferons, interleukins)
* Type 1 diabetes only: polyclonal regulatory T cell and/or dendritic cell therapy
* Bleeding disorder
* Women of childbearing potential: Pregnant/ nursing (Note: Eligibility may be deferred per blood donation timelines for pregnancy/nursing)
* Diabetic patients only: Any clinical condition that might be adversely affected by the removal of up to 100 mL of blood
* An employee who is under the direct/ indirect supervision of the PI/ a co-investigator/ the study manager
* A direct study team member

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants from the clinic environment/ local providers/ diabetes events, relatives/ friends of participants, employees, and normal healthy participants from the community
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2026-06-09 (Estimated); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
Identification of circulating biomarkers that correlate with beta cell death in type 1 diabetes compared to healthy controls | Baseline
  The measure will be changes in beta cell death.
Changes in frequency of circulating biomarkers that correlate with beta cell death from type 1 diabetes patients compared to other cohorts | Baseline
  The measure will be changes in beta cell death.

CONTACTS AND LOCATIONS:
Overall Officials: Rupangi Vasavada, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: Undecided